CLINICAL TRIAL: NCT06077097
Title: Traumatic Events in Childhood, Attachment, Pain Perception, Epigenetic Marks, Quality of Life and Resilience: When Psychological Dimensions Interfere With the Hospital Management of Pain
Brief Title: Traumatic Events in Childhood, Attachment, Pain Perception, Epigenetic Marks, Quality of Life and Resilience.
Status: Completed | Type: Observational
Sponsor: University of Lorraine (Other)
Responsible Party: Principal Investigator, Christine Rotonda, Methodologist/Epidemiologist Head of Research Unit, Pierre Jane Centre, University of Lorraine
Other Study IDs: 2022-A02519-34
Record Dates: First submitted 2023-08-25; First posted 2023-10-11 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Chronic Pain; Adverse Childhood Experiences; Attachment Styles; Chronic Stress; Resilience, Psychological; Quality of Life; Epigenesis, Genetic
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — 1) measurement of cortisol levels 2) measurement of methylation of OXTR, NR3C1 and FKBP5 receptors and genes For the measurement of cortisol and methylation of the OXTR, NR3C1 and FKBP5 receptors and genes, blood cells will be collected, within the chronic pain structures, during the participant's inclusion visit if he/she agrees to participate in the biological ancillary study.
  The blood sample will be taken from the participant's fingertip by transcutaneous pricking, collecting a few drops of blood capillary. According to the recent study by Walker et al (98), DNA methylation profiles from dried blood spots are of good quality, strongly correlated with those of paired EDTA tube samples (mean r = 0.991).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Genetic: Biological samples — This project also includes an auxiliary exploratory biological study of subcellular mechanisms, using high-throughput sequencing (Next Generation Sequencing, NGS) to identify gene expression variations in order to determine the resilience/vulnerability of the variables studied with respect to the DC experience (cytogenetics and transcriptome).

SUMMARY:
In the present research study, aiming to explore the links between several psychological factors and chronic pain, the research seeks to develop an inclusive framework to investigate the role of adverse childhood experiences (ACEs) in patients' pain perception and overall quality of life throughout their pain management programs. Specifically, attachment styles (AS) and pain-related resilience processes are considered as potential mediators of the effectiveness of chronic pain management programs. Additionally, biological measures are proposed to investigate physiological parameters of pain and to further explore the degree of consistency between self-reported measures, ACEs, ASs, chronic stress, and several epigenetic biomarkers.

DETAILED DESCRIPTION:
One in four French adults suffers from chronic pain (CP), making it one of the main causes of long-term disability and disease burden in France. Despite the various pain management plans, which have brought their share of improvements, CP remains extremely resistant to treatment, and its annual health costs represent a major national problem. Considering that 70% of CP patients remain severely undertreated, managed exclusively by general practitioners and CP specialists, there is an emerging need to implement more effective and cost-efficient interdisciplinary pain management programs, following a biopsychosocial framework for the management of pain. This framework integrates biological, psychological, and social measures and their interactions to highlight an individual's unique pain state.

The psychological concept of "adverse childhood experiences" (ACEs) may play a role in the development and maintenance of CP. Researchers point to a frequency-dependent relationship between ACEs and chronic conditions in adulthood, with a higher number of ACEs leading to more severe CP problems in adulthood. However, research is still in its infancy, and it cannot be concluded that there is a causal relationship between ACEs and the development of persistent pain.

It is, therefore, essential to consider several factors that may potentially mediate this relationship, such as the psychological concept of adult attachment style. The latter refers to the way relationships with others are formed, shaped in early childhood. Attachment patterns can be characterized along two dimensions: attachment anxiety (worry about the availability of others) and attachment avoidance (discomfort with proximity and interdependence). Insecure attachment patterns (high anxiety and/or avoidance) have been associated with the development of chronic conditions such as fatigue, medically unexplained CP, and migraines. Furthermore, in patients with CP, attachment anxiety is associated with increased pain. Experimental pain studies have also shown a positive relationship between attachment anxiety and pain. In contrast, the results concerning attachment avoidance are contradictory. Attachment patterns are of great importance for the current project, as CP management programs are usually based on patient-to-patient talk groups, and the medical devices are occupied by doctors and carers. Therefore, the medical discourse, as well as the discourse of peers (i.e. other patients), will not have the same impact or importance depending on whether patients have developed secure attachments or not.

Based on the evidence presented above, it seems that the psychological constructs of ACEs and attachment may open up new avenues for understanding individual differences in the context of CP management programs. The research is particularly interested in complementing this line of reasoning by investigating individual differences in various epigenetic markers and levels of resilience of individuals to better understand how potentially traumatic life events will have different effects on patients and their treatment effectiveness.

The project aims to develop a more inclusive framework to study the role of ACEs in patients' pain perception and overall quality of life throughout their pain treatment, exploring the potential mediating effect of attachment styles, resilience, and deoxyribonucleic acid (DNA) methylation levels. The project is innovative in its assessment of multiple genetic receptors through the application of an ancillary biological study and in its application of a longitudinal research design.

ELIGIBILITY:
Inclusion Criteria:

* Have a chronic pain syndrome persisting for at least six months
* Have been referred to a chronic pain management programme at the Centre of evaluation and treatment of chronic pain at the "Belle- Isle" hospital (private hospital in Metz, France) or at the Pain Consultation of the Regional University Hospital of Nancy, France
* Be between 18 and 65 years old
* Be able to read and write in French (be able to understand the information and fill in the questionnaires independently)
* Agree to participate in the project and sign the consent form

Exclusion Criteria:

* Have received pain management in a specialised chronic pain facility (of any kind) during their lifetime
* Have physical, cognitive and/or linguistic deficiencies that make it impossible to fill in the questionnaires
* Have a psychiatric history (psychosis type)
* Have a drug or alcohol dependency
* Be a protected adult, under guardianship or curatorship
* Being pregnant or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The study population will consist of participants who have been diagnosed with a chronic pain syndrome for more than 6 months and who will be admitted for the first time to a hospital pain management programme in one of the regional structures specialised in the management of chronic pain (SDC), i.e. the Centre of Evaluation and Treatment of pain at the "Belle-Isle" hospital (private hospitals in Metz, France UNEOS Group) and the Pain Consultation of the Regional University Hospital (CHRU) at Nancy, France. Participants will be included for 12 months. All patients meeting the inclusion criteria and not meeting the non-inclusion criteria will be invited by the physicians performing the first consultation at the centres of inclusion to participate in the study before the start of any medical programme.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-04-12 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2024-12-18 (Actual)

PRIMARY OUTCOMES:
Observe the reported pain intensity and pain affect in individuals experiencing chronic pain | Baseline. Through study completion, an average of 1 year.
  Pain intensity and pain affect will be measured using the Numerical Rating Scale (NRS). The Numerical Rating Scale is typically an 11-point scale, with 0 representing "no pain" and 10 representing "the worst pain imaginable." In the case of pain intensity, higher scores on the NRS indicate worse pain, with 10 being the most severe pain. For pain affect, higher scores on the NRS may indicate more negative affective responses related to pain.

SECONDARY OUTCOMES:
Attachment Styles | Baseline. Through study completion, an average of 1 year.
  The different Attachment Styles (AS) will be identified using the Experiences in Close Relationships-Revised Questionnaire (ECR-R). It is a 36-item self-report questionnaire that assesses AS in romantic relationships. It consists of two dimensions: attachment anxiety and attachment avoidance. Participants rate each of the 36 statements using a 7-point likert scale which ranges from 1-strongly disagree to 7-strongly agree. Interpretation: Higher scores indicate a worse outcome in terms of attachment-related anxiety/avoidance, reflecting greater insecurity in romantic relationships.
Adverse childhood experiences | Baseline. Through study completion, an average of 1 year.
  The number of Adverse Childhood Experiences (ACEs) will be assessed using the Adverse Childhood Experiences International Questionnaire (ACE-IQ).
  The total number of ACEs to which the participant has been "exposed" is summed to create an ACE score ranging from 0 (no ACEs) to 13. A score of 0 ACEs means a low level of adversity and a score of 13 means a major level of adversity.
Assess the Quality of Life of individuals experiencing chronic pain | Baseline. Through study completion, an average of 1 year.
  Quality of life will be assessed using the SF-12 questionnaire. Two summary scores are reported from the SF-12 - a mental component score (MCS-12) and a physical component score (PCS-12). The scores may be reported as Z-scores (difference compared to the population average, measured in standard deviations). The United States population average PCS-12 and MCS-12 are both 50 points. The United States population standard deviation is 10 points. So each 10 increment of 10 points above or below 50, corresponds to one standard deviation away from the average. Higher scores on the SF-12 scale generally signify better physical and mental health, fewer limitations in daily activities, less pain, and a more positive perception of overall well-being. Conversely, lower scores suggest poorer health, more limitations, more pain, and a less positive perception of well-being.
Pain cognitions | Baseline. Through study completion, an average of 1 year.
  Pain cognitions, assessed using the Pain Beliefs and Perceptions Inventory (PBPI) The Pain Beliefs and Perceptions Inventory (PBPI) is a questionnaire comprising 16 items that assess individuals' beliefs about pain across four primary dimensions: mystery, permanence, constancy, and self-blame. Respondents rate each item on a 4-point scale, ranging from -2 (strongly disagree) to 2 (strongly agree). In summary, higher scores on these PBPI subscales reflect stronger beliefs and perceptions in the respective dimensions of pain. Interpretation of these scores should consider the context of the study and the specific research questions or hypotheses being investigated.
Pain Interference | Baseline. Through study completion, an average of 1 year.
  The impact of pain on daily behaviour, measured using the Concise Pain Questionnaire (CPQ). The questionnaire assesses the degree of pain interference in seven daily activities using a Likert scale from 0 (no interference) to 10 (complete interference). Higher scores indicate more significant pain-related disruption to these activities, while lower scores suggest minimal interference. A minimum of four completed items out of seven is required to calculate the mean pain interference score, offering a concise measure of pain's impact on daily life.
Pain resilience | Baseline. Through study completion, an average of 1 year.
  Pain resilience processes as measured by the Pain Resilience Scale modified version for chronic pain (PRS)
  This scale comprises 12 items and 2 factors measuring cognitive/affective positivity and behavioral perseverance respectively. Respondents rate their agreement with each item using a Likert scale ranging from 0 ("not at all") to 4 ("all the time").
  Higher scores in the cognitive/affective factor indicate a greater perceived ability to maintain cognitive and emotional positivity despite severe or prolonged pain.
  Higher scores in the behavioral perseverance factor indicate a greater perceived ability to persist in various behaviors even when faced with prolonged or severe pain.

OTHER OUTCOMES:
Epigenetic measurements related to childhood adversity | Baseline. Through study completion, an average of 1 year.
  The percentage of methylation of genes encoding the target regions of the OXTR receptor and the NR3C1 and FKBP5 genes from whole blood, saliva and oral cells, assessed by Methylated DNA Immunoprecipitation (MeDIP) assays in combination with PCR to map the location and determine the abundance of modified histones or variants in the genome.
Stress Measurement | Baseline. Through study completion, an average of 1 year
  Stress measurement: cortisol concentration in blood by enzyme immunoassay (EIA)

CONTACTS AND LOCATIONS:
Overall Officials: CYRIL CYRIL, Pr, Principal Investigator — UR 4360 APEMAC, UNIVERSITY OF LORRAINE
Locations (1):
- Ur 4360 Apemac, Metz, Lorraine,, France

IPD SHARING:
Plan to Share IPD: No